CLINICAL TRIAL: NCT00097799
Title: An Open Label, Non-randomized Treatment Protocol of Tipranavir Co-administered With Low-dose Ritonavir (TPV/r) in Protease Inhibitor-experienced Patients With HIV-1 Infection (the Tipranavir Expanded Access Program)
Brief Title: Tipranavir Expanded Access Program (EAP) in PI-experienced Patients With HIV-1 Infection
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1182.70
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

INTERVENTIONS:
Drug: Tipranavir — 500 mg twice daily
Drug: Ritonavir — 200 mg twice daily

SUMMARY:
This study was designed to provide early access to and evaluate the safety of TPV/r in PI-experienced patients with HIV-1 infection.

Age Groups: Child, Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (115):
- United States (115):
  - 1182.70.127 Health Services Center, Inc., Anniston, Alabama
  - 1182.70.006 Spectrum Medical Group, Phoenix, Arizona
  - 1182.70.016 Health for Life Clinic, Little Rock, Arkansas
  - 1182.70.065, Anaheim, California
  - 1182.70.246, Baldwin Park, California
  - 1182.70.043, Fountain Valley, California
  - 1182.70.092, Fresno, California
  - 1182.70.057, Glendale, California
  - 1182.70.064, Harbor City, California
  - 1182.70.079, Long Beach, California
  - 1182.70.015, Los Angeles, California
  - 1182.70.053, Los Angeles, California
  - 1182.70.066, Los Angeles, California
  - 1182.70.071, Los Angeles, California
  - 1182.70.137, Los Angeles, California
  - 1182.70.198, Los Angeles, California
  - 1182.70.008, Newport Beach, California
  - 1182.70.081, Oakland, California
  - 1182.70.095, Oakland, California
  - 1182.70.067, Panorama City, California
  - 1182.70.033, San Diego, California
  - 1182.70.014, San Francisco, California
  - 1182.70.020, San Francisco, California
  - 1182.70.048, San Francisco, California
  - 1182.70.085, San Francisco, California
  - 1182.70.214, San Francisco, California
  - 1182.70.022, San Rafael, California
  - 1182.70.222, Stanford, California
  - 1182.70.005, Tarzana, California
  - 1182.70.030, Tarzana, California
  - 1182.70.068, Woodland Hills, California
  - 1182.70.218 Denver Infectious Disease Consultants, Denver, Colorado
  - 1182.70.281, Denver, Colorado
  - 1182.70.074, New Haven, Connecticut
  - 1182.70.073, Norwich, Connecticut
  - 1182.70.032, Washington D.C., District of Columbia
  - 1182.70.042, Washington D.C., District of Columbia
  - 1182.70.289 Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - 1182.70.003, Fort Lauderdale, Florida
  - 1182.70.013, Fort Lauderdale, Florida
  - 1182.70.049, Fort Lauderdale, Florida
  - 1182.70.096, Fort Lauderdale, Florida
  - 1182.70.045, Fort Myers, Florida
  - 1182.70.026, Hollywood, Florida
  - 1182.70.023, Miami, Florida
  - 1182.70.040, North Palm Beach, Florida
  - 1182.70.007, Orlando, Florida
  - 1182.70.117, Plantation, Florida
  - 1182.70.017, Pompano Beach, Florida
  - 1182.70.047, West Palm Beach, Florida
  - 1182.70.002, Atlanta, Georgia
  - 1182.70.046, Atlanta, Georgia
  - 1182.70.069, Atlanta, Georgia
  - 1182.70.037, Dactur, Georgia
  - 1182.70.058, Jesup, Georgia
  - 1182.70.174, Macon, Georgia
  - 1182.70.019, Chicago, Illinois
  - 1182.70.029 Dr. David Moore, Chicago, Illinois
  - 1182.70.194, Chicago, Illinois
  - 1182.70.010, Joliet, Illinois
  - 1182.70.167, Indianapolis, Indiana
  - 1182.70.192, Iowa City, Iowa
  - 1182.70.099, New Orleans, Louisiana
  - 1182.70.025 Chase Brexton Health Services, Inc, Baltimore, Maryland
  - 1182.70.082, Boston, Massachusetts
  - 1182.70.090, Boston, Massachusetts
  - 1182.70.004, Berkley, Michigan
  - 1182.70.084, Detroit, Michigan
  - 1182.70.035, St Louis, Missouri
  - 1182.70.242, St Louis, Missouri
  - 1182.70.093, Lincoln, Nebraska
  - 1182.70.021, Las Vegas, Nevada
  - 1182.70.288 Hackensack University Medical Center, Hackensack, New Jersey
  - 1182.70.075, Sommers Point, New Jersey
  - 1182.70.024, Briarcliff Manor, New York
  - 1182.70.105, Bronk, New York
  - 1182.70.039, Kingston, New York
  - 1182.70.028, New York, New York
  - 1182.70.031, New York, New York
  - 1182.70.036, New York, New York
  - 1182.70.050, New York, New York
  - 1182.70.062, New York, New York
  - 1182.70.104, New York, New York
  - 1182.70.086 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 1182.70.250 Montefiore Medical Center, The Bronx, New York
  - 1182.70.061, Asheville, North Carolina
  - 1182.70.100, Chapel Hill, North Carolina
  - 1182.70.136 Mecklenburg Medical Group, P.A., Charlotte, North Carolina
  - 1182.70.103, Durham, North Carolina
  - 1182.70.241 University of CIncinnati Medical Center, Cincinnati, Ohio
  - 1182.70.044, Portland, Oregon
  - 1182.70.059 Fanno Creek Clinic, Portland, Oregon
  - 1182.70.077 Kaiser Permanente-IDC, Portland, Oregon
  - 1182.70.051, Philadelphia, Pennsylvania
  - 1182.70.080, Philadelphia, Pennsylvania
  - 1182.70.072, Providence, Rhode Island
  - 1182.70.126, Charleston, South Carolina
  - 1182.70.271, Charleston, South Carolina
  - 1182.70.088, Columbia, South Carolina
  - 1182.70.165 Comprehensive Care Center, Nashville, Tennessee
  - 1182.70.018, Austin, Texas
  - 1182.70.038, Dallas, Texas
  - 1182.70.041, Dallas, Texas
  - 1182.70.055, Dallas, Texas
  - 1182.70.070, Dallas, Texas
  - 1182.70.060, El Paso, Texas
  - 1182.70.052, Houston, Texas
  - 1182.70.054, Houston, Texas
  - 1182.70.285, Houston, Texas
  - 1182.70.128 Olmos Park Medical Associates, San Antonio, Texas
  - 1182.70.011, Annadale, Virginia
  - 1182.70.217, Richmond, Virginia
  - 1182.70.097, Seattle, Washington
  - 1182.70.76, Seattle, Washington
  - 1182.70.083, Spokane, Washington